CLINICAL TRIAL: NCT01027338
Title: Tai Chi Exercise in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Tai Chi Exercise in Patients With COPD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Russell Phillips, MD, Beth Israel Deaconess Medical Center
Other Study IDs: K24AT000589 (NIH)
Record Dates: First submitted 2009-12-04; First posted 2009-12-07 (Estimated); Last update posted 2009-12-07 (Estimated); Status verified 2009-12

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Aquatic Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tai Chi Exercise (Experimental)
  Interventions: Other: Tai chi exercise
- Usual Care (No Intervention)

INTERVENTIONS:
Other: Tai chi exercise
  Arms: Tai Chi Exercise

SUMMARY:
This is a pilot randomized controlled trial of feasibililty and prelimnary effects of a 12 week tai chi intervention vs. usual care in patients with chronic obstructive pulmonary disease

ELIGIBILITY:
Inclusion Criteria:

* physician diagnosis of COPD
* FEV1<65% of predicted and FEV1/FVC<70% of predicted
* ≥45 years old

Exclusion Criteria:

* COPD exacerbation requiring ER visit or hospitalization within past month
* planned major pulmonary intervention in coming 3 months
* severe peripheral vascular disease/claudication or other physical condition precluding walk test
* inability to perform bicycle ergometry
* severe cognitive dysfunction (MMSE ≤ 24)
* inability to speak English
* current participation in a pulmonary rehabilitation or regular practice of tai chi

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
study feasibility

SECONDARY OUTCOMES:
quality of life
exercise capacity

CONTACTS AND LOCATIONS:
Overall Officials: Gloria Y Yeh, MD, MPH, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States